CLINICAL TRIAL: NCT05345418
Title: Evaluation of the Safety and Efficacy of Umbilical Cord-Derived Mesenchymal Stem Cell (VCELL 1) for Male Patients With Sexual Deficiency: A Phase I/IIa Randomised Crossover Trial
Brief Title: Umbilical Cord-Derived Mesenchymal Stem Cell (VCELL 1) for Male Patients With Sexual Deficiency
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ISC.21.08
Record Dates: First submitted 2022-04-14; First posted 2022-04-25 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sexual Dysfunction Male
Keywords: Sexual Dysfunction Male; reproductive hormones; mesenchymal stem Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord-Derived Mesenchymal Stem Cell, then Placebo (group A) (Experimental): Cohort 1 will receive two single intravenous dose of UC MSCs of 1.5 million cells per kilogram body weight on their Study Month 0, and Study Month 3.
  - Each treatment period was separated by a 4 - week washout to allow the effective systemic elimination of the UC MSCs before subsequent treatment initiation
  Interventions: Biological: Umbilical Cord-Derived Mesenchymal Stem Cell for Male Patients with Sexual Deficiency
- Placebo, then Umbilical Cord-Derived Mesenchymal Stem Cell (group B) (Active Comparator): Cohort 2 will receive two single intravenous dose of UC MSCs of 1.5 million cells per kilogram body weight on their Study Month 7, and Study Month 10
  Interventions: Biological: Umbilical Cord-Derived Mesenchymal Stem Cell for Male Patients with Sexual Deficiency

INTERVENTIONS:
Biological: Umbilical Cord-Derived Mesenchymal Stem Cell for Male Patients with Sexual Deficiency — Patients will receive two administrations at a dose of 1.5 million cells/kg patient bodyweight via the IV route with a 3-month intervening interval. A validated umbilical cord blood mesenchymal stem cells (UC-MSC) line was selected from the Vinmec Tissue Bank and cultured under xeno-free, serum-free and antibiotic-free conditions as previously described. To prepare UC-MSCs for therapy, aliquots of Passage 3 (P3) UC-MSCs will be thawed and cultured to P5 to get approximately 500 million cells and dispensed to 10 million UC-MSCs/ml/vial for cryopreservation. Upon request from the clinical team, aliquots of P5 UC-MSCs will be thawed in a temperature control water bath or incubator on the infusion day. The UC-MSCs will be washed and suspended in Ringer Lactate.

SUMMARY:
Sexual functional deficiency affects largely the physical conditions, life and sexual quality of the patients. Hypogonadism affects about 4 to 5 million men in the US, and the incidence increases with age. In our recent phase I clinical trial, we have shown that intravenous adipose - derived MSC administration was safe in female and male patients with hormone deficiency. Post-transplantation sexual satisfaction was observed in all patients enrolled in this study. Testosterone levels in males increased significantly after transplantation and were maintained at high levels for up to 6 months before decreasing again at the 12-month follow-up. The aim of this clinical trial was to assess the safety and effectiveness of allogeneic administration of MSCs in middle-aged people with sexual functional deficiency.

DETAILED DESCRIPTION:
Sexual functional deficiency occurs at some point in life and becomes a problematic issue in middle-aged adulthood. Regenerative medicine, especially mesenchymal stem cell (MSC) transplantation, has developed extensively, with preclinical and clinical trials emphasizing the benefits of stem cell therapy for restoration of sexual deficiency. n our recent phase I clinical trial, we have shown that intravenous adipose - derived MSC administration was safe in female and male patients with hormone deficiency. Post-transplantation sexual satisfaction was observed in all patients enrolled in this study. Testosterone levels in males increased significantly after transplantation and were maintained at high levels for up to 6 months before decreasing again at the 12-month follow-up. The aim of this clinical trial was to assess the safety and effectiveness of allogeneic administration of MSCs in middle-aged people with sexual functional deficiency. In phase II, 40 males with hormone deficiency will be recruited and divided randomly into two groups (n=23 each). The group A will receive UC-MSCs intravenously at day 0 and day 90 ± 7, while the group B will be infused with UC-MSCs at day 180 ± 14 and day 270 ± 14. Each group will be monitored for 365 ± 14 days after the first infusion. The phase II is to investigate safety and efficacy of UC-MSC infusion for the treatment of sexual hormone deficiency in males.

The primary outcome are: (1) numbers of AEs or SAEs during UC-MSC infusion and 365 ± 14 days after the first infusion; (2) Testosterone levels and sexual life quality through quantification of Aging Men Symptom (AMS), International Index of Erectile Function (IIEF), and Sexual Quality of Life Questionnaire (SQoL-M) at day 90 ± 7 and day 180 ± 14 of the group A compared to those of the group B.

The secondary outcome are: (1) Testosterone levels and (2) sexual life quality through quantification of AMS, IIEF, and SQoL-M at day 90 ± 7, day 180 ± 14, and day 365 ± 14 after the first UC-MSC infusion of each group compared to the baseline; (3) cytokine concentration (TNFa, IFN-γ, IL1, IL-6, IL-8, IL-4, IL-10, IDO) in serum of the participants and their T cell immunophenotype at day 90 ± 7, day 180 ± 14, and day 365 ± 14 after the first UC-MSC infusion.

ELIGIBILITY:
Inclusion Criteria:

* Males with sexual hormone deficiency aged 50 to 70 years
* AMS score ≥ 27
* IIEF < 14
* SQoL-M ≤ 87
* and Testosterone ≤ 12 nMol/L
* Normal liver function (ALT, AST and Bilirubin are normal according to biological index of Vietnamese people).
* Normal kidney function is usually according to the biological index of Vietnamese people.
* No infection, HIV, HBV, active syphilis.
* Must provide written informed consent.

Exclusion Criteria:

* The patient had surgery to remove the gonads.
* Patients with a history of cancer, or undergoing cancer treatment, or are positive for cancer screening tests including: PSA, AFP, Pepsinogen I, Pepsinogen II and erythrocyte smear test.

The patient is taking anti-rejection drugs.

* Patients with malformations, malformations or tumors of the endocrine glands.
* Endocrine impairment due to diabetes (HBA1c > 7) and other metabolic diseases.
* Patients with active autoimmune disease or positive for antinuclear antibodies.
* Patients with severe heart failure, severe renal failure, severe liver failure, severe respiratory failure, history of cerebral infarction, myocardial infarction, Alzeimer.
* Patients with hypothyroidism.
* The patient has an acute infection.
* Patients with clinically significant coagulopathy or other hematological diseases.
* History of allergy to anesthetics, anesthetics, antibiotics.
* Patients who are using other hormone-improving drugs or supplements (including Sildenafil) in the last 2 weeks or want to continue using these drugs during the study period.
* The patient is a smoker.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males with sexual hormone deficiency
Enrollment: 158 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The safety of allogenic umbilical cord-derived mesenchymal stem cell administration for the treatment of hormone deficiency in male | up to the 12-month period following treatment
  To assess safety, the number of AEs or SAEs during stem cell administration up to the 12-month period following treatment will be evaluated
Testosterone levels | up to the 12-month period following treatment
  To evaluate the Testosterone levels of the patients with sexual functional deficiency
Changes in sexual life quality using Aging Men Symptom (AMS) | up to the 12-month period following treatment
  AMS includes 10 items
Changes in sexual life quality through quantification of International Index of Erectile Function (IIEF) | up to the 12-month period following treatment
  IIEF includes 15 items
Changes in sexual life quality through quantification of Sexual Quality of Life Questionnaire (SQoL-M) | up to the 12-month period following treatment
  IIEF includes 11 items

CONTACTS AND LOCATIONS:
Overall Officials: Tan Sinh Nguyen, Dr, Principal Investigator — Vinmec Times City International Hospitalme
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang ZY, Xing XY, Ju GQ, Zhong L, Sun J. Mesenchymal stem cells from human umbilical cord ameliorate testicular dysfunction in a male rat hypogonadism model. Asian J Androl. 2017 Sep-Oct;19(5):543-547. doi: 10.4103/1008-682X.186186. PMID 27586027
- [Background] Kouchakian MR, Baghban N, Moniri SF, Baghban M, Bakhshalizadeh S, Najafzadeh V, Safaei Z, Izanlou S, Khoradmehr A, Nabipour I, Shirazi R, Tamadon A. The Clinical Trials of Mesenchymal Stromal Cells Therapy. Stem Cells Int. 2021 Nov 3;2021:1634782. doi: 10.1155/2021/1634782. eCollection 2021. PMID 34745268
- [Background] Kadihasanoglu M, Ozbek E. Mesenchymal stem cell therapy in treatment of erectile dysfunction: Autologous or allogeneic cell sources? Int J Urol. 2016 Apr;23(4):348-9. doi: 10.1111/iju.13058. Epub 2016 Jan 28. No abstract available. PMID 26822742